CLINICAL TRIAL: NCT01846858
Title: Histological Characterization of Vaginal Cuff Tissue Using Different Energy Sources During Robotic Hysterectomy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rosanne M. Kho, M.D., Associate Professor of Obstetrics-Gynecology, Mayo Clinic
Other Study IDs: 10-001538
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Extent of Thermal Injury Using Different Energy Sources at the Time of Robotic Hysterectomy Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10 vaginal tissue specimens from each group of energy modality will be compared and analyzed. Tissue from the specimen side of the hysterectomy will be sent (after marking the most distal edge with a marker) for pathological evaluation such that the vaginal length is not compromised.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CO2 Laser
- Monopolar energy

SUMMARY:
Vaginal cuff dehiscence, a rare complication of gynecologic surgeries, can be devastating, particularly when associated with bowel evisceration. A review of records from 1970 - 2001 at the Mayo Clinic in Rochester, MN revealed a low incidence (0.032%) of vaginal cuff dehiscence after pelvic operation via both abdominal and vaginal approaches3. At a single, large, tertiary care facility, total laparoscopic hysterectomy (TLH) was associated with an increased incidence of vaginal cuff dehiscence compared to other approaches (4.93% vs. 0.29% TVH, and 0.12% TAH)1. A review of our robotic experience revealed a vaginal cuff dehiscence incidence of 4.1%, which is comparable to the previously reported incidence for TLH2. An increasing number of laparoscopic hysterectomies are being performed in the United States with the rate of laparoscopic procedures increasing from 0.3% in 1990 to 11.8% in 20034. With 11.8% of 600,000 annual hysterectomies being performed via the laparoscopic route in the United States, there would be an estimated 3,400 cases of vaginal cuff dehiscence per year.

The cause of the higher rate of vaginal cuff dehiscence in both laparoscopic and robotic hysterectomies is currently unknown. One of the major differences between the laparoscopic and robotic approach as compared to the vaginal/abdominal route is the method by which the cervix is amputated from the vagina. With the vaginal and abdominal approaches, a colpotomy is made sharply with a knife or scissors. In contrast, the colpotomy is performed with electrocoagulation with the laparoscopic and robotic routes. One theory to explain the increased dehiscence incidence is the lateral thermal effects of electrocoagulation on the vaginal cuff which may adversely affect tissue healing.

This study aims primarily to shed light on the etiology of vaginal cuff healing after a robotic total hysterectomy. This will be done by comparing the extent of thermal injury at the cellular level using monopolar vs CO2 laser at the time of the colpotomy.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Patient over age of 18 years undergoing a robotic total hysterectomy
* Patients in Mayo Clinic (Arizona)

Exclusion Criteria:

* Patients with gynecologic malignancy involving the vagina

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for a robotic hysterectomy for benign indications
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Extent of thermal injust grossly from free tissue edge (mm) | at 12 and 6 o'clock

CONTACTS AND LOCATIONS:
Overall Officials: Rosanne M Kho, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States